CLINICAL TRIAL: NCT04652167
Title: What is the Diagnostic and Prognostic Accuracy of C-reactive Protein, Serum Procalcitonin and Soluble Urokinase Plasminogen Activator Receptor in the Initial Investigation of Patients With Suspected Community-acquired Pneumonia
Brief Title: Diagnostic Accuracy of Infection Biomarkers in the Initial Investigation of Patients With Suspected Pneumonia
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-11d-2020
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pneumonia, Bacterial
Keywords: C-reactive protein,; serum procalcitonin,; soluble urokinase plasminogen activator receptor
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected of community-acquired pneumonia: All patients admitted to the emergency department with suspected community- acquired pneumonia by the attending physician
  Interventions: Diagnostic Test: PCT; Diagnostic Test: suPAR; Diagnostic Test: Standard care

INTERVENTIONS:
Diagnostic Test: PCT — Serum PCT concentration is quantified with an automated sandwich immunoassay "ECLIA" (Elecsys®, BRAHMS PCT-analyses) on Cobas e801. Calibration (BRAHMS PCT LIA assay) is performed once per reagent lot and no later than 24 h after Cobas e pack has been registered in the instrument. Quality control is performed after each calibration.
Diagnostic Test: suPAR — Serum suPAR was measured using suPARnostic© Turbilatex assay reagents (validated on Cobas© c111) protocol for Cobas© c702 and c502 applying the Multi-Pack cassettes (Roche Diagnostics, Mannheim, Germany). Calibration is performed at least once a month or in connection to a new batch of TurbiLatex reagents, after calibration a quality control is performed.
Diagnostic Test: Standard care — Standard care is the measurement of CRP (C-reactive protein) will be measured with C - reactive protein (CRP4) immunoturbidimetric assay (Tina-quant®, Roche) on Roche/Hitachi cobas© systems c701/702. Calibration is performed (Tina-quant® C - reactive protein IV) once per reagent lot and after 6 months using the same reagent lot. Quality control is required after calibration and according manufacturing instructions.

SUMMARY:
The aim of this study is to investigate the diagnostic and prognostic value of C-reactive protein (CRP), serum procalcitonin (PCT) and soluble urokinase plasminogen activator receptor (suPAR) in the initial investigation of patients acute hospitalized with suspected community-acquired-pneumonia (CAP)

DETAILED DESCRIPTION:
Target pneumonia treatment should be initiated within a few hours, which is why early and accurate diagnosis is extremely important. Uncertain or delayed diagnosis will often lead to an overconsumption of broad-spectrum antibiotics, which contributes to increased development of resistant bacteria and thus threaten the treatment options of the future. Pneumonia diagnosis is primarily made today on the basis of clinical symptoms and findings in the form of cough, vomiting, chest pain, fever, shortness of breath, supplemented with X-ray of the lungs, relevant blood tests and analysis of expectoration. However, X-ray is an imprecise diagnostic tool. The diagnosis of CAP is challenged by nonspecific symptoms, uncertain diagnostic methods and waiting time for test results up to several days.

Therefore, numerous studies have investigated biomarkers that can possibly support the diagnosis of CAP. C-reactive protein (CRP) and serum procalcitonin (PCT) are biomarkers that may distinguish CAP from other causes of acute respiratory infections. The CRP biomarker has been endorsed as a guide for antibiotic treatment by the National Institute for Health and Care Excellence (NICE) and PCT was suggested by the American Infectious Diseases Society of America. Soluble urokinase plasminogen activator receptor (suPAR) has emerged as a potentially novel biomarker for inflammatory diseases including pneumonia. Several studies have highlighted suPAR as a significant prognostic mortality marker and strongly related to disease severity and worse outcome in a variety of conditions. It is also a promising biological marker in the diagnosis of CAP.

The diagnostic value of the optimal biomarkers for the diagnosis of CAP remains controversial. The investigators hypothesize that serum CRP, PTC and suPAR have an impact on diagnosing, prognosis, and treatment of patients with a verified community-acquired-pneumonia. The objectives of the study are:

* To identify the diagnostic accuracy of CRP, PCT and suPAR in community-acquired pneumonia
* To identify the prognostic value of CRP, PCT and suPAR in relation to adverse events

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Patients suspected with pneumonia by the attending physician. The physician will base his/her suspicion on e.g. clinical symptoms such as cough, increased sputum production, chest tightness, dyspnea and fever > 38⁰C, and indication for chest x-ray

Exclusion Criteria:

* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted at the emergency department with suspected pneumonia by the attending physician.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic of community acquired pneumonia | expert assessment within 3 months after patient discharge from the hospital
  The percentage of patients diagnosed with community-acquired pneumonia determined by an expert panel. This outcome measure is a binary variable - verified pneumonia or no pneumonia.
  The expert panel consists of two independent consultants from the emergency department with experience in infection and emergency medicine, who individually will determine whether the patient admitted with suspected community-acquired pneumonia, had the diagnosis. The diagnosis will be based on all available relevant information from the patient medical record within 48 hours from admission including computed tomography. A standardized template will be used. Disagreement will be discussed until a consensus is reached.
  .

SECONDARY OUTCOMES:
Intensive care unit (ICU) treatment | within 60 days from admission to the emergency department
  Transfer to the intensive care unit will be recorded during the current hospitalization as a binary variable (transferred/not-transferred)
Length of hospital stay (LOS | within 60 days from current admission to the emergency department
  Defined as the time (in days) spent in hospital during the current admission. Measured in days from admission to hospital discharge. Discharge date minus admission date.
30-days mortality | 30 days from the admission to the emergency department
  Mortality within 30 days from admission to the Emergency Department
90-days mortality | 90 days from the admission to the emergency department
  Mortality within 90 days from admission to the Emergency Department
Readmission | within 30 days from the discharge to the hospital
  If a subject is admitted over a 30 day period after the current hospitalization discharge measured as a binary outcome Re-admissions/not re-admissions
In-hospital mortality | within 60 days from admission to the emergency department
  Patient mortality during the current hospitalization. Binary outcome - Died/ Not died

OTHER OUTCOMES:
CURB-65 score for predicting mortality in community-acquired-pneumonia: | within 4 hours from admission
  CURB-65 score consists of: Confusion of new onset, Blood Urea nitrogen greater than 7 mmol/L (19 mg/dL), respiratory rate of 30 breaths per minute or greater, blood pressure less than 90 mmHg systolic or diastolic blood pressure 60 mmHg or less and age 65 or older. The score stratify patients to groups 1 (mild pneumonia), 2 (moderate pneumonia) and 3-5 (severe pneumonia).
Pneumonia severity index (PSI): | within 4 hours from admission
  Risk classes to predict the severity of pneumonia. Scores are given based on demographics, comorbidity, clinical measurements and physical Exam Findings (<70 = Risk Class II, 71-90 = Risk Class III, 91-130 = Risk Class IV, >130 = Risk Class V)
Microbial agents | results within 7 days from sputum sample collection
  Microbial agents (bacteria and viruses) identified in standard culture, PCR and multiplex PCR. Sputum samples are collected within 1 hour from patient admission.
  Descriptive findings in percentage will be registered
Level of markers of lung injury | within 4 hours from admission
  serum surfactant protein D, KL-6 and YKL-40

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Chair — University Hospital of Southern Denmark
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnstone J, Mandell L. Guidelines and quality measures: do they improve outcomes of patients with community-acquired pneumonia? Infect Dis Clin North Am. 2013 Mar;27(1):71-86. doi: 10.1016/j.idc.2012.11.001. PMID 23398866
- [Background] Musher DM, Thorner AR. Community-acquired pneumonia. N Engl J Med. 2014 Oct 23;371(17):1619-28. doi: 10.1056/NEJMra1312885. No abstract available. PMID 25337751
- [Background] Hey J, Thompson-Leduc P, Kirson NY, Zimmer L, Wilkins D, Rice B, Iankova I, Krause A, Schonfeld SA, DeBrase CR, Bozzette S, Schuetz P. Procalcitonin guidance in patients with lower respiratory tract infections: a systematic review and meta-analysis. Clin Chem Lab Med. 2018 Jul 26;56(8):1200-1209. doi: 10.1515/cclm-2018-0126. PMID 29715176
- [Background] Wussler D, Kozhuharov N, Tavares Oliveira M, Bossa A, Sabti Z, Nowak A, Murray K, du Fay de Lavallaz J, Badertscher P, Twerenbold R, Shrestha S, Flores D, Nestelberger T, Walter J, Boeddinghaus J, Zimmermann T, Koechlin L, von Eckardstein A, Breidthardt T, Mueller C. Clinical Utility of Procalcitonin in the Diagnosis of Pneumonia. Clin Chem. 2019 Dec;65(12):1532-1542. doi: 10.1373/clinchem.2019.306787. Epub 2019 Oct 15. PMID 31615771
- [Background] Loonen AJM, Kesarsing C, Kusters R, Hilbink M, Wever PC, van den Brule AJC. High pneumococcal DNA load, procalcitonin and suPAR levels correlate to severe disease development in patients with pneumococcal pneumonia. Eur J Clin Microbiol Infect Dis. 2017 Sep;36(9):1541-1547. doi: 10.1007/s10096-017-2963-2. Epub 2017 Mar 29. PMID 28353184
- [Background] Ni W, Han Y, Zhao J, Cui J, Wang K, Wang R, Liu Y. Serum soluble urokinase-type plasminogen activator receptor as a biological marker of bacterial infection in adults: a systematic review and meta-analysis. Sci Rep. 2016 Dec 19;6:39481. doi: 10.1038/srep39481. PMID 27991579
- [Background] Song S, Jia Q, Chen X, Lei Z, He X, Leng Z, Chen S. Serum suPAR associated with disease severity and mortality in elderly patients with community-acquired pneumonia. Scand J Clin Lab Invest. 2020 Oct;80(6):515-522. doi: 10.1080/00365513.2020.1795920. Epub 2020 Jul 27. PMID 32716662
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497